CLINICAL TRIAL: NCT01124370
Title: Safety and Efficacy Evaluation of Respicardia Therapy for Central Sleep Apnea
Brief Title: Chronic Evaluation of Respicardia Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Respicardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Respicardia - Chronic Study I
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Sleep Disordered Breathing; Cheyne Stokes Respiration; Periodic Breathing; Sleep Apnea; Central Sleep Apnea
Keywords: Sleep Disordered Breathing; Cheyne Stokes Respiration; Periodic Breathing; Sleep Apnea; Central Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Cheyne-Stokes Respiration; Sleep Apnea, Central | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): All enrolled subjects will undergo attempted system implantation and therapeutic assessment. Subjects' baseline assessment values will serve as control parameters for the therapy evaluation.
  Interventions: Device: remedē (TM) system

INTERVENTIONS:
Device: remedē (TM) system — Implantation of the remedē (TM) system, including implantable pulse generator, stimulation lead, and (optional) sensing lead. Nightly provision of unilateral transvenous phrenic nerve therapy during sleep periods.
  Other Names: Respicardia Therapy; Cardiac Concepts Therapy; (note: Respicardia was formerly Cardiac Concepts)

SUMMARY:
The purpose of this study is to determine the chronic safety and efficacy of phrenic nerve stimulation on central sleep apnea (CSA). Clinically, CSA events translate into sleep fragmentation, excessive daytime sleepiness, reduced exercise capacity, and possibly ventricular arrhythmias.

The study is chronic in nature, such that subjects will undergo the implantation of an implantable pulse generator and stimulation lead. A sensing lead may also be placed during the initial implant procedure. Subjects will be followed for up to six-months on therapy to assess respiratory and heart failure outcomes. Following the six-month therapy visit, subjects will enter into a long-term follow-up phase until the completion of the study.

It is anticipated that data obtained in this study will show that the proposed intervention can modify respiration with a low incidence of adverse effects. The results of this trial are intended to be used to develop a subsequent protocol for pivotal study.

ELIGIBILITY:
Inclusion Criteria:

* Candidate is at least 18 years old
* Candidates with known recent history of Periodic Breathing, as evidenced by an overnight polysomnogram (PSG) within 60 days of the implant procedure demonstrating:

  * Apnea-Hypopnea Index (AHI) greater than or equal to 20 events/hr
  * Predominantly central origin (central apnea events comprise 50% or more of all apnea events)
  * Limited obstructive events (obstructive apneas comprise less than 20% of the AHI)

Exclusion Criteria:

* Candidates who are pregnant
* Candidates with baseline oxygen saturation less than or equal to 90% on a stable FiO2
* Candidates with severe COPD
* Candidates with a history of cerebrovascular accident (CVA), myocardial infarction, coronary artery bypass grafting (CABG) surgery, or percutaneous coronary intervention (PCI) within the 3 months prior to the study
* Candidates with unstable angina
* Candidates with history of primary pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Ponikowski, MD, Principal Investigator — 4th Military Clinical Hospital with Polyclinic, Poland; William T Abraham, MD, Principal Investigator — Ohio State University
Locations (13):
- United States (5):
  - BryanLGH Heart Institute, Lincoln, Nebraska
  - The Ohio State University, Columbus, Ohio
  - Lancaster Heart and Stroke Foundation, Lancaster, Pennsylvania
  - St. Thomas Heart, Nashville, Tennessee
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
- Germany (4):
  - Heart and Diabetes Center, Bad Oeynhausen
  - Köln University, Cologne
  - University of Kiel, Kiel
  - St. Adolf-Stift Hospital, Reinbek
- Policlinico di Monza-IRCCS, Monza, Italy
- Poland (3):
  - Jagiellonian University, Krakow
  - Medical Military Institute, Warsaw
  - 4th Military Hospital, Wroclaw

REFERENCES:
- [Derived] Javaheri S, McKane SW, Cameron N, Germany RE, Malhotra A. In patients with heart failure the burden of central sleep apnea increases in the late sleep hours. Sleep. 2019 Jan 1;42(1):zsy195. doi: 10.1093/sleep/zsy195. PMID 30325462
- [Derived] Abraham WT, Jagielski D, Oldenburg O, Augostini R, Krueger S, Kolodziej A, Gutleben KJ, Khayat R, Merliss A, Harsch MR, Holcomb RG, Javaheri S, Ponikowski P; remede Pilot Study Investigators. Phrenic nerve stimulation for the treatment of central sleep apnea. JACC Heart Fail. 2015 May;3(5):360-369. doi: 10.1016/j.jchf.2014.12.013. Epub 2015 Mar 11. PMID 25770408

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Implantation of the remedē system which provides unilateral transvenous phrenic nerve stimulation therapy during sleep.
Period: Overall Study
Arm/Group | Treatment
Started | 57 (Underwent implant attempt)
Successfully Implanted | 50
Therapy Initiated | 48
3 Month Visit | 47 (Defines evaluable population)
Completed | 37 (Completed 2 year post-implant follow-up)
Not Completed | 20

BASELINE CHARACTERISTICS:
Population: All subjects with an implant attempt.
Arm/Group | Treatment
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 51
Region of Enrollment [Number; unit: participants]
  United States | 19
  Poland | 17
  Germany | 18
  Italy | 3
Apnea-Hypopnea Index (AHI) [Mean (Standard Deviation); unit: events/hour] — The number of apneas and hypopneas per hour of sleep. An apnea is defined by 3 characteristics:
  1. There is a drop in the peak thermal sensor excursion or alternate nasal air pressure transducer (inspiratory effort) by > 90% of baseline
  2. The duration of the event lasts at least 10 seconds
  3. At least 90% of the event's duration meets the amplitude reduction criteria for apnea
  Hypopnea defined as 30% reduction in airflow (or alternative hypopnea sensor) for ≥10 seconds over at least 90% of the event's duration that is associated with a >4% fall in oxygen saturation from baseline
  events/hour | 49.1 (15.0)
Epworth Sleepiness Scale (ESS) [Mean (Standard Deviation); unit: units on a scale] — The ESS is an assessment to measure a subject's general level of daytime sleepiness. Scores can range from 0-24, with higher scores indicating higher level of daytime sleepiness.
  units on a scale | 8.6 (4.4)
Minnesota Living with Heart Failure Questionnaire (MNLHF) [Mean (Standard Deviation); unit: units on a scale] — This questionnaire was for the N=46 patients diagnosed with heart failure. Scores can range from 0-105, with lower scores indicating better quality of life.
  units on a scale | 41.4 (18.9)
Six minute hall walk [Mean (Standard Deviation); unit: meters] — N=55 subjects completed this assessment at baseline.
  meters | 377.8 (144.5)
New York Heart Association (NYHA) Functional Class [Number; unit: participants] — NYHA Class definitions:
  Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea Class II:Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV: Unable to carry on any physical activity without discomfort. Symptoms of HF at rest. If any physical activity is undertaken, discomfort increases.
  participants
    Not applicable | 11
    Class I | 4
    Class II | 28
    Class III | 13
    Class IV | 1
Heart failure [Number; unit: participants]
  Yes | 46
  No | 11
Ejection Fraction [Mean (Standard Deviation); unit: percent] — Available for N=54 participants.
  percent | 29.6 (10.8)
Coronary Artery Disease [Number; unit: participants]
  Yes | 35
  No | 22
Hypertension [Number; unit: participants]
  Yes | 41
  No | 16
Hyperlipidemia [Number; unit: participants]
  Yes | 20
  No | 37
Atrial Fibrillation [Number; unit: participants]
  Yes | 16
  No | 41
Concomitant implantable device delivering therapy [Number; unit: participants]
  Yes | 29
  No | 28

OUTCOME MEASURES:

1. Primary Outcome: AHI Change From Baseline at 3 Months
Description: Change = Month 3 score - Baseline score The Apnea-Hypopnea Index (AHI) is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep.
Time Frame: Baseline and 3 months on therapy
Population: The evaluable population includes subjects who completed a 3 Month post therapy initiation visit.
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Treatment
Number analyzed (Participants) | 47
events/hour | -27.1 (17.7)
Statistical Analysis 1: Comparison: Treatment; The null hypothesis was that there would be no change in AHI from baseline; Test type: Superiority or Other; p < .001, t-test, 2 sided — The test was conducted using a 0.05 level of significance

2. Secondary Outcome: Related Adverse Events
Description: The number of subjects with a serious adverse event (SAE) considered related to the remedē system or implant procedure is provided. The number of subjects with a non-SAE related to the remedē system or implant procedure is also provided. Events are included if they occurred on or after the initial implant date through 2 years post implant. A subject may have both SAE and non-SAE events, so the participants with serious events cannot be added to the non-serious participants to get the total number of participants experiencing a related event.
Time Frame: Up to 2 years
Population: Subjects with an implant attempt.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 57
participants
  Serious | 18
  Non-Serious | 23

3. Secondary Outcome: Epworth Sleepiness Scale Change From Baseline at 6 Months
Description: Change = Month 6 score - Baseline score The ESS is an assessment to measure a subject's general level of daytime sleepiness. Scores can range from 0-24, with higher scores indicating higher level of daytime sleepiness.
Time Frame: Baseline and 6 months on therapy
Population: Subjects with baseline and 6 month data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 46
units on a scale | -2.0 (4.3)

4. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire Change From Baseline at 6 Months
Description: Change = Month 6 score - Baseline score This questionnaire was for the N=46 patients diagnosed with heart failure. Scores can range from 0-105, with lower scores indicating better quality of life.
Time Frame: Baseline and 6 months on therapy
Population: Heart failure subjects with baseline and 6 month results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 36
units on a scale | -9.9 (16.5)

5. Secondary Outcome: Heart Failure Clinical Composite
Description: The composite is determined according to the following definitions.
  Worsened: subject died; was hospitalized due to or associated with worsening HF; demonstrated worsening in NYHA class at last observation carried forward; moderate-marked worsening of patient global assessment score at last observation carried forward; or permanently discontinued therapy from the remedē System due to or associated with worsening HF.
  Improved: subject did not worsen (as defined above) and demonstrated improvement in NYHA class at last observation carried forward or moderate-marked improvement in patient global assessment score at last observation carried forward.
  Unchanged: patient was neither improved nor worsened.
Time Frame: 6 months on therapy
Population: Evaluable subjects with heart failure at baseline.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 37
participants
  Improved | 20
  Unchanged | 9
  Worsened | 8

6. Secondary Outcome: Six-minute Hall Walk Test Change From Baseline at 6 Months
Description: Change = Month 6 score - Baseline score
Time Frame: Baseline and 6 months on therapy
Population: Subjects with baseline and 6 month data.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treatment
Number analyzed (Participants) | 39
meters | -7.5 (58.7)

7. Secondary Outcome: NYHA Functional Class Improvement From Baseline to 6 Months
Description: Shift in NYHA Class from baseline to 6 months NYHA Class I - Patients with cardiac disease but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea or anginal pain.
  NYHA Class II - Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea or anginal pain.
  NYHA Class III - Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea or anginal pain.
  NYHA Class IV - Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present event at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: Baseline and 6 months on therapy
Population: Heart failure subjects with 6 month data.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 36
participants
  Improved | 11
  No change | 25
  Worsened | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Events are included if they occurred on or after the initial implant date through 2 years post implant.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 41/57
Other Adverse Events (participants affected / at risk) | 35/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=57)
ACUTE CONGESTIVE HEART FAILURE (Cardiac disorders) | 14
LEAD DISLODGEMENT (General disorders) | 11
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 6
ACUTE CORONARY SYNDROME (Cardiac disorders) | 3
ATRIAL ARRHYTHMIA (Cardiac disorders) | 2
CHEST PAIN (Cardiac disorders) | 2
CORONARY ARTERY DISEASE (Cardiac disorders) | 2
CLOSTRIDIAL ENTERITIS (Gastrointestinal disorders) | 2
EXTRA-RESPIRATORY STIMULATION (General disorders) | 2
LEAD COMPONENT FAILURE (General disorders) | 2
BRONCHITIS (Infections and infestations) | 2
PNEUMONIA (Infections and infestations) | 2
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2
FRACTURE (Musculoskeletal and connective tissue disorders) | 2
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
STROKE (Nervous system disorders) | 2
URINARY TRACT INFECTION (Renal and urinary disorders) | 2
THROMBOSIS (Vascular disorders) | 2
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1
AV BLOCK (Cardiac disorders) | 1
HYPERTHYROIDISM (Endocrine disorders) | 1
DETACHED RETINA (Eye disorders) | 1
WORSENING OF CATARACTS (Eye disorders) | 1
GASTROENTERITIS (Gastrointestinal disorders) | 1
GI BLEEDING (Gastrointestinal disorders) | 1
HERNIA REPAIR (General disorders) | 1
IMPENDING POCKET PERFORATION (General disorders) | 1
INADEQUATE LEAD POSITION (General disorders) | 1
LOSS OF STIMULATION (General disorders) | 1
ATYPICAL PNEUMONIA (Infections and infestations) | 1
DIABETES (Metabolism and nutrition disorders) | 1
HYPEROSMOLAR SYNDROME (Metabolism and nutrition disorders) | 1
ATYPICAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
GOUT ATTACK (Musculoskeletal and connective tissue disorders) | 1
SPINAL CANAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1
HEAD AND NECK CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
EPILEPTIC SEIZURE (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 1
MENINGIOMA (Nervous system disorders) | 1
DELUSIONAL SYNDROME (Psychiatric disorders) | 1
RENAL DYSFUNCTION (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
COPD EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 1
PULMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
VOCAL CORD LESION (Respiratory, thoracic and mediastinal disorders) | 1
ATOPIC ECZEMA (Skin and subcutaneous tissue disorders) | 1
CRT-D DEVICE REPLACEMENT (Surgical and medical procedures) | 1
DEVICE EXPLANTATION (Surgical and medical procedures) | 1
HEMATOMA (Vascular disorders) | 1
HYPOTENSION (Vascular disorders) | 1
PERIPHERAL VASCULAR DISEASE (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=57)
DIAPHRAGMATIC STIMULATION DISCOMFORT (General disorders) | 16
URINARY TRACT INFECTION (Renal and urinary disorders) | 6
ACUTE CONGESTIVE HEART FAILURE (Cardiac disorders) | 3
EXTRA-RESPIRATORY STIMULATION (General disorders) | 3
PAIN (General disorders) | 3
HEMATOMA (Vascular disorders) | 3
HYPOTENSION (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No